CLINICAL TRIAL: NCT04115436
Title: Association of Genetic Variants With Risk of Stroke in Patients With Atrial Fibrillation Off-anticoagulation
Acronym: GSAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCAI_Natale
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Thromboembolic Events
Keywords: LAA isolation, stroke, anticoagulation
MeSH Terms: conditions — Thromboembolism; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stroke (+): Patients experiencing thromboembolic events following a brief discontinuation of anticoagulant or having thrombus on the LAA occlusion device
- No-stroke: Patients remaining stroke-free months after discontinuation of anticoagulants

SUMMARY:
Life-long therapy with oral anticoagulants (OAC) is strongly recommended in AF patients receiving left atrial appendage isolation (LAAI) to prevent thromboembolic (TE) events. However, some patients are observed to remain stroke-free while off OACs for years whereas others experience TE events if OAC is discontinued even for a short period of time. Therefore, we aim to evaluate the association of genetic variants (single nucleotide polymorphisms - SNPs) with off-anticoagulation stroke-risk in AF patients.

DETAILED DESCRIPTION:
1. BACKGROUND Atrial fibrillation (AF) is known to be a leading cause of thrombo-embolic (TE) events (1).The left atrial appendage (LAA), an embryological remnant of the primitive left atrium, has been reported to be the source of thrombus formation in more than 90% of patients with non-valvular AF (2). More specifically, the loss of contractile function in the LAA following electrical isolation of the appendage (LAAI) leads to stasis and thrombus formation, which may then embolize into the systemic circulation. For this reason, life-long oral anticoagulation (OAC) is strongly recommended in post-LAAI cases to reduce the stroke-risk. However, intolerance to OAC, non-compliance, increase in the risk of bleeding in patients with bleeding disorders or in elderly with high fall-risk and difficulty in maintaining the therapeutic level for certain novel oral anticoagulants in patients with renal dysfunction are several limitations of the OAC therapy (3). Furthermore, patients occasionally need to discontinue OACs as advised by their treating physicians while undergoing other medical procedures. Patient-preference and non-compliance are other important reasons for OAC discontinuation.

   Whatever may be the cause, the consequence in terms of TE events, is observed to be highly variable. Some patients experience a TE event after withdrawal of OAC for a very short period while others remain stroke-free even after years while off OAC therapy. This intriguing observation triggers a vital question; does genetics play a role in increasing predisposition to stroke or providing protection from TE events? The current pilot study aims to address that question as understanding the underlying molecular mechanism would be highly useful in risk-prediction, counselling and optimal management of post-LAAI patients.

   Prior studies have reported an association between several single-nucleotide polymorphisms (SNPs) with stroke in patients with or without AF (4-19). Most were documented to be linked with elevated stroke-risk whereas few were found to have a protective impact. However, SNPs associated with stroke in the post-LAAI cases have not been elucidated yet. More importantly, it is not known why discontinuation of OAC has a differential impact on this high-risk population. Therefore, in this pilot study, we aim to test a number of SNPS (a list is provided at the end of the protocol) in post-LAAI cases to determine their association with stroke after discontinuation of OAC.

   1.1 Safety This study poses minimal risk to the subject. More specifically, the risks are those that are associated with venipuncture (pain, bleeding, bruising, infection, and inflammation at the site), during the single blood specimen collection.
2. STUDY RATIONALE We hypothesize that there will be significant differences in the allele frequencies of SNPs among patients with and without TE events.
3. STUDY OBJECTIVES 3.1 Primary Objective To compare the SNP profile of post-LAAI patients that have or have not experienced any TE events after discontinuation of OAC.
4. STUDY DESIGN 4.1 Study Overview This is a single center, observational clinical trial. Subjects who meet all inclusion criteria and none of the exclusion criteria will be screened and consecutive consenting patients will be enrolled in the study. We will screen all patients that have stopped OAC after LAAI and enroll the consenting patients that have or have not experienced stroke during discontinuation of OAC.

The total duration of subject participation will be 1 day. The total duration of the study is expected to be 1 year.

ELIGIBILITY:
Inclusion Criteria:

- i. male or female over 18 years of age at the time of enrollment ii. have received LAAI procedure iii. Discontinued OAC for any duration

Exclusion Criteria:

* i. end-stage renal or liver disease ii. on oral anticoagulation for any other condition iii. pregnant, breastfeeding, or unwilling to provide consent iv. presence of other conditions or abnormalities that in the opinion of the Investigator would compromise the quality of the data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: AF patients following LAA isolation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of difference in the SNP profile between the Stroke (+) and no-stroke patients | 1 day
  Proportion of difference in the SNP profile between the Stroke (+) and no-stroke patients

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Cardiac Arrhythmia Institute, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No